CLINICAL TRIAL: NCT03555708
Title: Mobility Exercises for Gait (MEG Neuroplasticity Project)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0082-18-FB; Department Funding (Other Grant/Funding Number: Munroe Meyer Institute)
Record Dates: First submitted 2018-05-11; First posted 2018-06-13 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy
Keywords: Gait Training; Power Training; Action-Perception Training; Brain Imaging; Mobility
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Velocity Power Training (Experimental): Training will consist of unilateral and bilateral leg presses (Total Gym GTS, San Diego CA), which will primarily target the quadriceps followed by the hip extensors and plantarflexors. Target load will be 40% to 80% of 1-repetition maximum (1RM) with progression toward 80%. Each participant will perform 3 to 5 sub-maximal efforts followed by 6 sets of 5 maximum-effort repetitions at the predetermined percentage of 1RM for each leg separately. Following the unilateral leg presses, 6 sets of 5 repetitions of bilateral leg presses will be performed at the predetermined percentage of 1RM. To minimize fatigue, 1-2 minutes of rest will be given between sets.
  Interventions: Other: Physical Therapy
- Perception-Action Physical Therapy (Experimental): The therapy includes: activities of adequate intensity that promote gait adaptation and gait speed sustainment, exploratory activities that enhance the somatosensory experience through rich/novel movement, and optimally challenging activities that emphasize planning and problem solving that requires altering the leg kinematics to meet the environmental and task constraints. This includes a 15-minutes of sustaining and adapting gait speed while walking along a 40-meter hallway. Participants will alter their gait through exploratory movements. During the following 20 minutes participants will perform discrete problem solving activities including: waling backward sand stair negotiation.
  Interventions: Other: Physical Therapy
- Body Weight Supported Treadmill Training (Experimental): The child will walk on the treadmill for 35-minutes, while the body weight is supported with an overhead system at 30 percent of the child's body weight, reducing every other week by 10 percent until no support is provided during the final 2 weeks. Treadmill speed will be set at 90% of the child's over ground walking speed, gradually increasing each session. Speed adjustments depend on the child's ability to control their steps and achieve: activities that promote symmetry of the leg kinematics, activities that promote maintaining an upright lower limb posture and clearing the tow during the swing, and activities that promote pushing off with ankle at terminal stance.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Physical therapy will be implemented three times a week with subjects over an eight week span. Each physical therapy session will last 40-minutes and will be conducted by a licensed physical therapist.
  Other Names: Therapeutic Gait Training

SUMMARY:
This study is directed at identifying a the neurophysiological changes seen in children with cerebral palsy (CP) after undergoing physical therapy. The specific aims of the study will: (1) determine the changes in the sensorimotor cortical activity after physical therapy, (2) determine the mobility, participation and muscular performance improvements after therapy, and (3) determine the changes in a child's participation in activities outside of the laboratory environment.

DETAILED DESCRIPTION:
This study is directed at identifying a the neurophysiological changes seen in children with cerebral palsy (CP) after undergoing physical therapy. The specific aims of the study will: (1) determine the changes in the sensorimotor cortical activity after physical therapy, (2) determine the mobility, participation and muscular performance improvements after therapy, and (3) determine the changes in a child's participation in activities outside of the laboratory environment. The study consists of a cohort of children with CP that will undergo an action-perception training protocol, a cohort that will undergo a high velocity power training protocol and a cohort that will undergo body weight supported treadmill training. Participants will be between the ages of 9-18 years and have gross motor function classification score levels between I-III. All participants will complete final initial baseline measures of their brain activity, mobility, muscle performance, and participation activity outside of the laboratory. After completing these tests, the children will undergo the respective physical therapy protocols for 8-weeks (3 days a week). After the 8-weeks of therapy, both groups will repeat the same tests that were completed at baseline. Follow-up assessment will consist of a physical therapist scheduling a time to visit the family at their house and ask them questions about the child's participation in activities.

ELIGIBILITY:
Inclusion Criteria:

* Sustained a brain injury around the time of birth or a diagnosis of Cerebral Palsy
* Must be able walk without a wheelchair (GMFCS I-III)

Exclusion Criteria:

* Children dependent on a wheel chair for mobility
* Braces, permanent retainers, or metal in the head (creates artifact in the MEG)
* Orthopedic surgery within last 6 months
* Botulinum injections within the last 6 months

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Brain Activity in Motor Cortices - MEG | Baseline and 8 weeks
  To assess the activity of the motor cortices, the child will produce an isometric knee extension force to match a target that is between 5-30% of his/her maximum voluntary force. The children will be instructed to perform the target matching task as rapidly and as accurately as possible. The MEG experiment will involve the child performing ~120 isometric target matching trials.
Change in Brain Activity in Sensory Cortices - MEG | Baseline and 8 weeks
  To assess the activity of the somatosensory cortices, a tactile stimulation will be applied to the bottom of the foot at the first metatarsal using a small airbladder. For each child, 120 paired-pulse trials will be collected using an inter-stimulus interval of 500 ms, and an inter-pair interval that randomly varied between 4.5 and 4.8 s.
Change in Mobility - 10-Meter Walk | Baseline and 8 weeks
  The childs 10-meter preferred and fast-as-possible walking speeds will be evaluated. The children will complete three trials at each speed, and the mean of the respective trials will be the key metric. During these tests, the child will walk across a GaitRITE digital mat (CIR Systems, Sparta, NJ) that will quantify the walking speed, step length, step width and cadence.
Change in Mobility - 1-Minute Walk | Baseline and 8 weeks
  The child's walking endurance will be assessed by asking them to walk as far as possible for a one-minute time period. Cones will be placed at the ends of a 40-m hallway and the child will be asked to walk back and forth during the time period. During the walk the child will wear a heart-rate monitor and wireless accelerometers that are positioned on the lower back and feet. The heart-rate monitor will be used as an indirect measure of the child's physical fitness, while the accelerometers will be used assess the child's dynamic balance.

SECONDARY OUTCOMES:
Change in Resting Cortical Activity - MEG | Baseline and 8 weeks
  The resting state activity of the brain will also be collected. This will involve the child sitting quietly with his/her eyes closed for 5 minutes.
Change in Mobility - Dynamic Gait Index | Baseline and 8 weeks
  The child will be asked to perform a series of mobility tasks such as stepping over shoe-box, changing their gait speed, walking up stairs, turning head while walking, etc. These series of standardized test will be used to assess the child's gait adaptability.
Change in Muscle Performance - Biodex | Baseline and 8 weeks
  A Biodex System 3 dynamometer will be used to assess the isometric strength and power production of the right and left knee joint musculature separately. Standard alignment of the knee joint axis with the dynamometer and set-up will be implemented. Separate knee extensor and flexor isometric strength tests will initially be measured from three maximal trials with the knee flexed at 90 degrees. This will be followed by the child performing maximal knee extensor/flexion concentric contractions with the dynamometer set at 30 deg/sec, 60 deg/sec and 120 deg/sec. The peak torque generated from the five contractions performed in each of the respective sets will be used as an outcome variable.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline and 3 Months Post and 6 Months Post Treatment
  Survey that evaluates the child's self-reported physical activity, strength and pain. The PROMIS will be completed at baseline and at the 3 and 6 months after therapy. A physical therapist will perform the 3 and 6 month follow-up assessments at the family's home.
Change in Participation in Environment Measure for Children and Youth (PEM-CY) | Baseline and 3 Months Post and 6 Months Post Treatment
  A survey to be completed by the child's parent/primary caregiver to gather information about the child's current level of participation in home, school and community environments. The survey will provide information regarding frequency of various activities performed, level of involvement during these activities and the parent/caregivers level of desire to see change in the child's involvement in activities. The PEM-CY will be completed at baseline and at the 3 and 6 months after therapy. A physical therapist will perform the 3 and 6 month follow-up assessments at the family's home.
Change in Activity - Actograph | Baseline 2 week days and two weekends, Post Treatment 2 week days and two weekends
  The child will wear an activity tracker at their waist while they are at home, in the community and at school. The activity tracker will be worn for 2 weekdays and 2 weekend days. The average across this time period will be used to assess the activity levels of the child outside of the laboratory setting. These measurements will be performed at baseline and after completing the therapy protocol
Change in Hoffmann Reflex (H-reflex) | Baseline and 8 weeks
  This tests is similar to how a medical doctor performs a tendon tap to assess a child's reflexes. The only difference is the methods that will be employed in this study can quantify the magnitude of the reflex. The H-reflex will be elicited by simulating the tibial or median nerve with a constant current electrical simulator. the muscular activity generated by the stimulus will be measured with EMG. The peak amplitude of the H-reflex seen in the EMG signal will be determined by gradually increasing the stimulus until the amplitude of the reflex no longer increases. Changes in the amplitude before the therapy and after will be used as an indirect assessment of spinal cord plasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Max J Kurz, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center Munroe Meyer Institute, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI and all of the investigators have made a commitment to publish, in a timely manner, all of the relevant scientific information that they will derive during this project. Publications will be in accordance with NIH guidelines. Unpublished information will be made available to interested parties via a request to the Principal Investigator (Dr. Kurz). Following publication, raw neuroimaging (MEG, MRI), biomechanical data, and clinical assessments will be made publicly available to the research community through a hyperlink on the PI's personal website at the University of Nebraska Medical Center (UNMC). These data will be de-identified, in accordance with the rules of the Institutional Review Board (IRB) of the UNMC. Such data sharing will allow replication of this study's primary findings, as well as opportunities for new findings as other investigators may apply different analysis methods, including new methods that may emerge in the future.
Supporting Information: Study Protocol, CSR
Time Frame: Upon completion of study and data analysis.
Access Criteria: Contact Dr. Kurz